CLINICAL TRIAL: NCT03043066
Title: The Effect of Non-surgical Periodontal Therapy With or Without Systemic Administration of Amoxicillin and Metronidazole on Serum Levels of TRAP-5b in Patients With Generalized Chronic Periodontitis - A Comparative Clinical Study
Brief Title: Serum TRAP-5b Levels in Patients With Generalized Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MADC/IRB-IX/2016/193
Record Dates: First submitted 2017-01-28; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; TRAP-5b; Non-surgical periodontal therapy; Systemic antibiotics
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Group A - scaling and root planing Group B - scaling and root planing along with antibiotic intervention of amoxicillin and metronidazole
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A -control group (Placebo Comparator): 15 subjects underwent scaling and root planing
  Interventions: Procedure: Scaling and root planing
- Group B-Interventional group (Active Comparator): 15 subjects underwent scaling and root planing along with antibiotic intervention of amoxicillin of 500 mg and metronidazole of 400 mg thrice daily for 7 days
  Interventions: Drug: scaling and root planing along with antibiotic intervention

INTERVENTIONS:
Procedure: Scaling and root planing — subjects underwent full mouth supragingival and subgingival scaling
  Other Names: Non-surgical periodontal therapy
  Arms: Group A -control group
Drug: scaling and root planing along with antibiotic intervention — subjects underwent full mouth supragingival and subgingival scaling along with antibiotic intervention of amoxicillin of 500 mg and metronidazole of 400 mg thrice daily for 7 days
  Other Names: Systemic antibiotics
  Arms: Group B-Interventional group

SUMMARY:
To compare the effect of non-surgical periodontal therapy with or without systemic administration of amoxicillin and metronidazole on the concentration of serum levels of TRAP-5b in patients with generalized chronic periodontitis.

DETAILED DESCRIPTION:
30 Chronic periodontitis subjects were divided into two groups- group A underwent scaling and root planing and group B underwent scaling and root planing with systemic administration of amoxicillin of 500 mg and metronidazole of 400 mg thrice daily for 7 days.

Periodontal parameters probing pocket depth and clinical attachment level were measured at baseline and at 3rd month. Serum TRAP-5b levels were also measured at baseline, 1 month and at 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* Presence of atleast 20 teeth
* more than 30% of sites with clinical attachment loss of ≥ 5 mm
* non-smokers
* no previous history of periodontal therapy

Exclusion Criteria:

* systemic diseases
* under antibiotics or anti-inflammatory drugs within previous 3 months
* pregnant and lactating women
* allergic to antibiotics

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Serum levels of TRAP-5b | Baseline and 3 months
  Concentration of serum levels of TRAP-5b was assessed at baseline and at 3rd month using ELISA method.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 3 months
  Probing pocket depth was measured using Williams periodontal probe at baseline and at 3rd month
Clinical attachment level | Baseline and 3 months
  Clinical attachment level was measured as a distance between base of pocket and a fixed point on the crown, such as cemento-enamel junction at baseline and at 3rd month.

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya CH, BDS, Principal Investigator — Meenakshi Ammal Dental College & Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosgarea R, Juncar R, Heumann C, Tristiu R, Lascu L, Arweiler N, Stavropoulos A, Sculean A. Non-surgical periodontal treatment in conjunction with 3 or 7 days systemic administration of amoxicillin and metronidazole in severe chronic periodontitis patients. A placebo-controlled randomized clinical study. J Clin Periodontol. 2016 Sep;43(9):767-77. doi: 10.1111/jcpe.12559. Epub 2016 Jun 23. PMID 27027501
- [Background] Keestra JA, Grosjean I, Coucke W, Quirynen M, Teughels W. Non-surgical periodontal therapy with systemic antibiotics in patients with untreated chronic periodontitis: a systematic review and meta-analysis. J Periodontal Res. 2015 Jun;50(3):294-314. doi: 10.1111/jre.12221. Epub 2014 Aug 21. PMID 25142259